CLINICAL TRIAL: NCT02175225
Title: Study of Deferoxamine Mesylate in Intracerebral Hemorrhage
Brief Title: Intracerebral Hemorrhage Deferoxamine Trial - iDEF Ttrial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Medical University of South Carolina (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Massachusetts General Hospital (Other); University of Massachusetts, Worcester (Other); University of Pennsylvania (Other); Johns Hopkins University (Other); Duke University (Other); University of North Carolina (Other); University of Florida (Other); Henry Ford Hospital (Other); Ohio State University (Other); St. Joseph's Hospital and Medical Center, Phoenix (Other); University of California, San Francisco (Other); Oregon Health and Science University (Other); Yale New Haven Health System Center for Healthcare Solutions (Other); University of Iowa (Other); Hartford Hospital (Other); The University of Texas Health Science Center, Houston (Other); Rhode Island Hospital (Other); Stanford University (Other); University of Washington (Other); University of Calgary (Other); Hopital de l'Enfant-Jesus (Other); University of Alberta (Other); Rush University Medical Center (Other); University Hospitals Cleveland Medical Center (Other); Columbia University (Other); Weill Medical College of Cornell University (Other); NYU Langone Health (Other); Mount Sinai Hospital, New York (Other); Loyola University (Other)
Responsible Party: Principal Investigator, Magdy Selim, MD, PhD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P000005; U01NS074425 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: Brain hemorrhage; Cerebral hemorrhage; Bleeding in the brain; Deferoxamine; iDEF trial
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages | interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deferoxamine Mesylate (Experimental): Deferoxamine Mesylate (32 mg/kg/day) given by an intravenous infusion for 3 consecutive days
  Interventions: Drug: Deferoxamine Mesylate
- Normal Saline (Placebo Comparator): Normal saline (0.9% sodium chloride) given by intravenous infusion for 3 consecutive days
  Interventions: Drug: Placebo (for Deferoxamine Mesylate)

INTERVENTIONS:
Drug: Deferoxamine Mesylate
  Arms: Deferoxamine Mesylate
Drug: Placebo (for Deferoxamine Mesylate)
  Arms: Normal Saline

SUMMARY:
The investigators hypothesize that treatment with the iron chelator, Deferoxamine Mesylate, improves the outcome of patients with brain hemorrhage.

The purpose of this study is to determine whether treatment with Deferoxamine Mesylate is of sufficient promise to improve outcome before pursuing a larger clinical trial to examine its effectiveness as a treatment for intracerebral hemorrhage.

DETAILED DESCRIPTION:
This is a prospective, multi-center, double-blind, randomized, placebo-controlled, phase-II clinical trial.

Subjects will be randomized to either deferoxamine mesylate (DFO) at 32 mg/kg/day (up to a maximum daily dose of 6000 mg/day), or saline placebo, given by IV infusion for 3 consecutive days.

Treatment will be initiated within 24 hours after ICH symptom onset. Randomization will control baseline imbalances associated with baseline ICH score, ICH onset-to-treatment time (OTT), ICH volume, baseline NIHSS score, and warfarin use.

All subjects will be followed for 6 months and will receive standard of care therapy while participating in the study.

Throughout the study, we will continue to assess the safety of DFO. At the conclusion of the study, the proportion of DFO-treated subjects with a good clinical outcome at 3 months (defined as modified Rankin Scale (mRS) score of 0-2) will be compared to the placebo proportion in a futility analysis to determine if it is futile to move DFO forward to Phase III efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years
* The diagnosis of ICH is confirmed by brain CT scan
* NIHSS score ≥6 and GCS >6 upon presentation
* The first dose of the study drug is expected to be administered within 24h of ICH symptom onset
* Functional independence prior to ICH, defined as pre-ICH mRS ≤1
* Signed and dated informed consent is obtained.

Exclusion Criteria:

* Previous chelation therapy or known hypersensitivity to DFO products
* Known severe iron deficiency anemia (defined as hemoglobin concentration < 7g/dL or requiring blood transfusions)
* Abnormal renal function, defined as serum creatinine >2 mg/dL
* Planned surgical evacuation of ICH prior to administration of study drug (placement of a catheter for ventricular drainage is not a contraindication to enrollment)
* SUSPECTED secondary ICH related to tumour, ruptured aneurysm or arteriovenous malformation, hemorrhagic transformation of an ischemic infarct, or venous sinus thrombosis
* Infratentorial hemorrhage
* Irreversibly impaired brainstem function (bilateral fixed and dilated pupils and extensor motor posturing)
* Complete unconsciousness, defined as a score of 3 on item 1a of the NIHSS (Responds only with reflex motor or autonomic effects or totally unresponsive, and flaccid)
* Pre-existing disability, defined as pre-ICH mRS ≥2
* Coagulopathy - defined as elevated aPTT or INR >1.3 upon presentation; concurrent use of direct thrombin inhibitors (such as dabigatran), direct factor Xa inhibitors (such as rivaroxaban or apixaban), or low-molecular-weight heparin
* Patients with confirmed aspiration, pneumonia, or evident bilateral pulmonary infiltrates on chest x-ray or CT scan prior to enrollment
* Patients with significant respiratory disease such as chronic obstructive pulmonary disease, pulmonary fibrosis, or any use (chronic or intermittent) of inhaled O2 at home
* FiO2 >0.35 (>4 L/min) prior to enrollment
* Sepsis (present source of infection ± lactic acidosis); Systemic Inflammatory Response Syndrome (Temp >100.4F or <96.8F; Heart rate >90; Respiratory rate >20 or PaCo2 <32 mmHg; WBC >12, <4, or bands >10%); or shock (SBP <90 mmHg) at presentation
* The presence of 4 or more of the following risk modifiers for ARDS prior to enrollment:

  1. Tachypnea (respiratory rate >30)
  2. SpO2 <95%
  3. Obesity (BMI >30)
  4. Acidosis (pH <7.35)
  5. Hypoalbuminemia (albumin <3.5 g/dL)
  6. Concurrent use of chemotherapy
* Taking iron supplements containing ≥ 325 mg of ferrous iron, or prochlorperazine
* Patients with heart failure taking > 500 mg of vitamin C daily
* Known severe hearing loss
* Known pregnancy, or positive pregnancy test, or breastfeeding
* Positive drug screen for cocaine upon presentation
* Patients known or suspected of not being able to comply with the study protocol due to alcoholism, drug dependency, noncompliance, living in another state or any other cause
* Any condition which, in the judgement of the investigator, might increase the risk to the patient
* Life expectancy of less than 90 days due to co-morbid conditions
* Concurrent participation in another research protocol for investigation of another experimental therapy
* Indication that a new DNR or Comfort Measures Only (CMO) order will be implemented within the first 72 hours of hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Selim, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (28):
- United States (25):
  - St. Joseph's Hospital / Barrow Neurological Institute, Phoenix, Arizona
  - Stanford University Medical Center, Palo Alto, California
  - San Francisco General Hospital, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Jacksonville, Florida
  - Loyola University Medical Center, Chicago, Illinois
  - RUSH University Medical Center, Chicago, Illinois
  - University of Iowa Medical Center, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Case Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University Medical Center, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Sciences Center, Houston, Texas
- Canada (3):
  - Foothills Hospital - University of Calgary, Calgary, Alberta
  - University of Alberta - Mackenzie Health Sciences Centre, Edmonton, Alberta
  - CHU de Québec - Hôpital de l'Enfant-Jésus, Québec

REFERENCES:
- [Background] Yeatts SD, Palesch YY, Moy CS, Selim M. High dose deferoxamine in intracerebral hemorrhage (HI-DEF) trial: rationale, design, and methods. Neurocrit Care. 2013 Oct;19(2):257-66. doi: 10.1007/s12028-013-9861-y. PMID 23943316
- [Background] Selim M, Yeatts S, Goldstein JN, Gomes J, Greenberg S, Morgenstern LB, Schlaug G, Torbey M, Waldman B, Xi G, Palesch Y; Deferoxamine Mesylate in Intracerebral Hemorrhage Investigators. Safety and tolerability of deferoxamine mesylate in patients with acute intracerebral hemorrhage. Stroke. 2011 Nov;42(11):3067-74. doi: 10.1161/STROKEAHA.111.617589. Epub 2011 Aug 25. PMID 21868742
- [Background] Selim M. Deferoxamine mesylate: a new hope for intracerebral hemorrhage: from bench to clinical trials. Stroke. 2009 Mar;40(3 Suppl):S90-1. doi: 10.1161/STROKEAHA.108.533125. Epub 2008 Dec 8. PMID 19064798
- [Background] Hatakeyama T, Okauchi M, Hua Y, Keep RF, Xi G. Deferoxamine reduces neuronal death and hematoma lysis after intracerebral hemorrhage in aged rats. Transl Stroke Res. 2013 Oct;4(5):546-53. doi: 10.1007/s12975-013-0270-5. PMID 24187595
- [Background] Xie Q, Gu Y, Hua Y, Liu W, Keep RF, Xi G. Deferoxamine attenuates white matter injury in a piglet intracerebral hemorrhage model. Stroke. 2014 Jan;45(1):290-2. doi: 10.1161/STROKEAHA.113.003033. Epub 2013 Oct 30. PMID 24172580
- [Background] Okauchi M, Hua Y, Keep RF, Morgenstern LB, Schallert T, Xi G. Deferoxamine treatment for intracerebral hemorrhage in aged rats: therapeutic time window and optimal duration. Stroke. 2010 Feb;41(2):375-82. doi: 10.1161/STROKEAHA.109.569830. Epub 2009 Dec 31. PMID 20044521
- [Background] Sonni S, Lioutas VA, Selim MH. New avenues for treatment of intracranial hemorrhage. Curr Treat Options Cardiovasc Med. 2014 Jan;16(1):277. doi: 10.1007/s11936-013-0277-y. PMID 24366522
- [Derived] Polymeris AA, Lioutas VA, Incontri D, Soman S, Selim MH; i-DEF Investigators. Evolution of Perihematomal Edema Mean Hounsfield Unit and Its Association with Clinical Outcome in Intracerebral Hemorrhage: A Post Hoc Analysis of the i-DEF Trial. Neurocrit Care. 2025 Dec;43(3):824-833. doi: 10.1007/s12028-025-02337-7. Epub 2025 Aug 11. PMID 40789806
- [Derived] Polymeris AA, Lioutas VA, Marchina S, Seiffge DJ, Roh DJ, Poyraz FC, Selim MH; i-DEF Investigators. Hemoglobin and Perihematomal Edema After Intracerebral Hemorrhage: A Post Hoc Analysis of the i-DEF Trial. Neurocrit Care. 2026 Feb;44(1):64-71. doi: 10.1007/s12028-025-02284-3. Epub 2025 May 21. PMID 40399657
- [Derived] Lee KH, Lioutas VA, Marchina S, Selim M; iDEF Investigators. The Prognostic Roles of Perihematomal Edema and Ventricular Size in Patients with Intracerebral Hemorrhage. Neurocrit Care. 2022 Oct;37(2):455-462. doi: 10.1007/s12028-022-01532-0. Epub 2022 Jun 8. PMID 35676589
- [Derived] Foster L, Robinson L, Yeatts SD, Conwit RA, Shehadah A, Lioutas V, Selim M; i-DEF Investigators. Effect of Deferoxamine on Trajectory of Recovery After Intracerebral Hemorrhage: A Post Hoc Analysis of the i-DEF Trial. Stroke. 2022 Jul;53(7):2204-2210. doi: 10.1161/STROKEAHA.121.037298. Epub 2022 Mar 21. PMID 35306827
- [Derived] Wei C, Wang J, Foster LD, Yeatts SD, Moy C, Mocco J, Selim M; i-DEF Investigators. Effect of Deferoxamine on Outcome According to Baseline Hematoma Volume: A Post Hoc Analysis of the i-DEF Trial. Stroke. 2022 Apr;53(4):1149-1156. doi: 10.1161/STROKEAHA.121.035421. Epub 2021 Nov 18. PMID 34789008
- [Derived] Lun R, Yogendrakumar V, Ramsay T, Shamy M, Fahed R, Selim MH, Dowlatshahi D. Predicting long-term outcomes in acute intracerebral haemorrhage using delayed prognostication scores. Stroke Vasc Neurol. 2021 Dec;6(4):536-541. doi: 10.1136/svn-2020-000656. Epub 2021 Mar 23. PMID 33758069
- [Derived] Selim M, Foster LD, Moy CS, Xi G, Hill MD, Morgenstern LB, Greenberg SM, James ML, Singh V, Clark WM, Norton C, Palesch YY, Yeatts SD; i-DEF Investigators. Deferoxamine mesylate in patients with intracerebral haemorrhage (i-DEF): a multicentre, randomised, placebo-controlled, double-blind phase 2 trial. Lancet Neurol. 2019 May;18(5):428-438. doi: 10.1016/S1474-4422(19)30069-9. Epub 2019 Mar 18. PMID 30898550

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferoxamine Mesylate: Deferoxamine Mesylate (32 mg/kg/day) given by an intravenous infusion for 3 consecutive days
  Deferoxamine Mesylate
- Normal Saline: Normal saline (0.9% sodium chloride) given by intravenous infusion for 3 consecutive days
  Placebo (for Deferoxamine Mesylate)
Period: Overall Study
Arm/Group | Deferoxamine Mesylate | Normal Saline
Started | 145 | 149
Initiated Study Drug | 144 (Subjects in whom study drug was not initiated are not subsequently followed per the protocol.) | 147 (Subjects in whom study drug was not initiated are not subsequently followed per the protocol.)
90 Day Outcome Obtained | 140 | 143
180 Day Outcome Obtained | 135 | 135
Completed | 137 | 138
Not Completed | 8 | 11
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 6 | 7
Not completed — Study drug not administered | 1 | 2

BASELINE CHARACTERISTICS:
Population: As specified in the Statistical Analysis Plan, the target population is the modified ITT population, including only subjects in whom study drug was initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferoxamine Mesylate | Normal Saline | Total
Number analyzed (Participants) | 144 | 147 | 291
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [51 to 71] | 62 [54 to 70] | 61 [52 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 112
  Male | 88 | 91 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 27 | 48
  Not Hispanic or Latino | 123 | 120 | 243
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 25 | 12 | 37
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 31 | 33 | 64
  White | 81 | 100 | 181
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Medical history: Hypertension [Count of Participants; unit: Participants] | 113 | 124 | 237
Medical history: Diabetes mellitus [Count of Participants; unit: Participants] | 32 | 43 | 75
Medical history: Cardiac disease [Count of Participants; unit: Participants] | 14 | 15 | 29
Medical history: Pulmonary disease [Count of Participants; unit: Participants] | 31 | 26 | 57
Medical history: Previous ischemic stroke or transient ischemic attack [Count of Participants; unit: Participants] | 10 | 16 | 26
Medical history: Previous intracerebral hemorrhage [Count of Participants; unit: Participants] | 7 | 3 | 10
Location of intracerebral hemorrhage [Count of Participants; unit: Participants]
  Lobar | 26 | 33 | 59
  Deep (thalamic) | 45 | 61 | 106
  Deep (non-thalamic) | 73 | 53 | 126
Intraventricular hemorrhage present [Count of Participants; unit: Participants] | 47 | 62 | 109

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Modified Rankin Scale (mRS) Score 0-2 at 90 Days
Description: The primary outcome measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-2 at 90 days. The mRS ranges from 0 to 6, with higher scores indicating worse outcome.
Time Frame: 90 days
Population: Per the SAP, the target population is the modified intention-to-treat population, including only subjects in whom study infusion is initiated. Complete case analysis was planned as the primary analytic approach.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 140 | 143
Participants | 48 | 47
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other — The alternative hypothesis, reflecting futility, is that the absolute treatment effect is less than 12% in favor of deferoxamine. In accordance with the futility design, futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference [AARD]); if the upper bound on the risk difference was less than 12% in favour of deferoxamine mesylate, this would be considered evidence of futility; Risk Difference (RD) = 0.006, 90% CI 1-sided [upper limit 0.068] — Futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference [AARD]); if UCB was less than 12% in favour of deferoxamine mesylate, this is considered evidence of futility

2. Primary Outcome: Number of Subjects Experiencing Serious Adverse Events
Description: Number of subjects experiencing Serious adverse events at any time from randomization through day 90
Time Frame: 90 days
Population: Per the SAP, the target population is the modified intention-to-treat population, including only subjects in whom study infusion is initiated.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 39 | 49
Statistical Analysis 1: Comparison: Deferoxamine Mesylate; Test type: Other; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.57 to 1.16]

3. Primary Outcome: Number of Subjects With Serious Adverse Events Within 7 Days
Description: Number of Subjects Experiencing Serious Adverse Events within 7 days of randomization
Time Frame: 7 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 24 | 26
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.57 to 1.56]

4. Secondary Outcome: Proportion of Patients With mRS Score 0-3 at 90 Days
Description: Another measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-3 at 90 days. The mRS ranges from 0 to 6, with higher scores indicating worse outcome.
  Although mRS 0-3 is less favorable than the primary outcome of mRS 0-2, it would still be a desirable effect in patients with ICH given that no treatments exist to reduce disability.
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 140 | 143
Participants | 91 | 82
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other — The alternative hypothesis, reflecting futility, is that the absolute treatment effect is less than 13% in favor of deferoxamine. In accordance with the futility design, futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference [AARD]); if the upper bound on the risk difference was less than13% in favor of deferoxamine mesylate, this would be considered evidence of futility; Risk Difference (RD) = 0.062, 90% CI 1-sided [upper limit 0.121] — Futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference[AARD]); if UCB was less than 12% in favour of deferoxamine mesylate, this is considered evidence of futility

5. Secondary Outcome: Proportion of Patients With Modified Rankin Scale (mRS) Score 0-2 at 180 Days
Description: Another measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-2 at 180 days. The mRS ranges from 0 to 6, with higher scores indicating worse outcome.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 135 | 135
Participants | 61 | 48
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 0.086, 90% CI 1-sided [upper limit 0.156] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Proportion of Patients With Modified Rankin Scale (mRS) Score 0-3 at 180 Days
Description: Another measure of efficacy is the modified Rankin Scale (mRS) score, dichotomized to define good functional outcome as mRS 0-3 at 180 days. The mRS ranges from 0 to 6, with higher scores indicating worse outcome.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 135 | 135
Participants | 97 | 92
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other — The alternative hypothesis, reflecting futility, is that the absolute treatment effect is less than 13% in favor of deferoxamine. In accordance with the futility design, futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference [AARD]); if the upper bound on the risk difference was less than 13% in favour of deferoxamine mesylate, this would be considered evidence of futility; Risk Difference (RD) = -0.018, 90% CI 1-sided [upper limit 0.029] — Futility was evaluated via the one-sided 90% upper confidence bound (90% UCB) of the treatment effect (absolute adjusted risk difference [AARD]); if UCB was less than 13% in favour of deferoxamine mesylate, this is considered evidence of futility

7. Secondary Outcome: Proportion of Subjects With Good Outcome (mRS 0-2) in the Early vs. Delayed Treatment Time Windows
Description: Analyses will be expanded to include an interaction between treatment and OTT window and the magnitude of the treatment effect, and corresponding confidence interval, will be estimated for each time window (<12 hours vs. >/= 12 hours) in order to explore the presence of a differential treatment effect in the OTT windows.
Time Frame: 90 days
Population: Per the SAP, the target population is the modified intention-to-treat population, including only subjects in whom study infusion is initiated. Complete case analysis was planned as the primary analytic approach. Subgroup analysis by Onset to treatment time window (<=12 hours vs >12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 140 | 143
Participants
  Onset to treatment time <=12 hours: number analyzed (Participants) | 42 | 46
  Onset to treatment time <=12 hours | 15 | 19
  Onset to treatment time >12 hours: number analyzed (Participants) | 98 | 97
  Onset to treatment time >12 hours | 33 | 28
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; p = 0.83, Regression, Logistic — The p value reflects the significance of the interaction term between treatment and onset to treatment time

8. Other Pre Specified Outcome: Ordinal Distribution of Scores on mRS at Day 90
Description: The overall ordinal distribution of scores on mRS at 90 days in DFO- and placebo-treated subjects will be determined.
Time Frame: 90 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 140 | 143
Participants
  mRS 0 | 6 | 4
  mRS 1 | 13 | 12
  mRS 2 | 29 | 31
  mRS 3 | 43 | 35
  mRS 4 | 33 | 43
  mRS 5 | 6 | 7
  mRS 6 | 10 | 11
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.72 to 1.67] — The estimation parameter is the adjusted common odds ratio

9. Other Pre Specified Outcome: Ordinal Distribution of Scores on mRS at 180 Days
Description: The overall ordinal distribution of scores on mRS at 180 days in DFO- and placebo-treated subjects will be determined.
Time Frame: 180 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 135 | 135
Participants
  mRS 0 | 10 | 5
  mRS 1 | 18 | 16
  mRS 2 | 33 | 27
  mRS 3 | 36 | 44
  mRS 4 | 22 | 24
  mRS 5 | 4 | 7
  mRS 6 | 12 | 12
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Odds Ratio, log = 1.26, 95% CI 2-sided [0.82 to 1.93]

10. Other Pre Specified Outcome: Adverse Event of Special Interest: Number of Patients With Allergic Reactions (During Infusion of Study Drug)
Description: Adverse event of special interest: anaphylaxis at any time during the study infusion
Time Frame: during the study infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 3 | 0

11. Other Pre Specified Outcome: Adverse Event of Special Interest: Number of Patients With Hypotension
Description: Hypotension requiring medical intervention at any time during the study infusion that could not be explained by other causes
Time Frame: during the study infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 1 | 2

12. Other Pre Specified Outcome: Adverse Event of Special Interest: Number of Patients With New Visual or Auditory Changes
Description: Adverse event of special interest: development of new and unexplained visual or auditory changes after initiation of the study infusion
Time Frame: after initiation of study infusion
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 3 | 4
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.0 to 14.97] — Confidence interval is exact (rather than asymptotic) due to small number of events

13. Other Pre Specified Outcome: Adverse Event of Special Interest: Number of Patients With Respiratory Compromise
Description: Adverse event of special interest: Respiratory compromise of any cause, including acute respiratory distress syndrome, in hospital until day 7 or discharge [whichever was earlier]
Time Frame: 7 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants
  All cause | 20 | 23
  Cause by acute respiratory distress syndrome | 2 | 1
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.51 to 1.54] — Confidence interval constructed only for all cause owing to small number of events caused by acute respiratory distress syndrome

14. Other Pre Specified Outcome: Number of Patients With Symptomatic Cerebral Edema
Description: Edema accompanied by an unexplained increase of more than four points on the US National Institutes of Health Stroke Scale or a decrease of more than two points in Glasgow Coma Scale score during the first week after the intracerebral haemorrhage.
Time Frame: 7 days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine Mesylate | Normal Saline
Number analyzed (Participants) | 144 | 147
Participants | 9 | 5
Statistical Analysis 1: Comparison: Deferoxamine Mesylate vs Normal Saline; Test type: Other; Risk Ratio (RR) = 1.84, 95% CI 2-sided [0.63 to 5.35]

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected until 180 days post-randomization. Serious adverse events were collected until 90 days post-randomization. Non-serious adverse events were collected until day 7 post-randomization or hospital discharge, whichever is earlier.
Description: Adverse events were classified with MedDRA v15 combined with Principal Investigator preferred adjustments.
Arm/Group | Deferoxamine Mesylate | Normal Saline
All-Cause Mortality (participants affected / at risk) | 12/144 | 12/147
Serious Adverse Events (participants affected / at risk) | 39/144 | 50/147
Other Adverse Events (participants affected / at risk) | 107/144 | 114/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine Mesylate (N=144) | Normal Saline (N=147)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound decomposition (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes increased (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Brain herniation (Nervous system disorders) | 4 (4) | 2 (2)
Brain midline shift (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 5 (5) | 2 (2)
CNS ventriculitis (Nervous system disorders) | 2 (2) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral hematoma expansion (Nervous system disorders) | 1 (1) | 2 (2)
Convulsion (Nervous system disorders) | 2 (2) | 1 (1)
Hydrocephalus (Nervous system disorders) | 4 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Neurological decompensation (Nervous system disorders) | 1 (2) | 4 (4)
Syncope/Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Withdrawal of life support (Surgical and medical procedures) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine Mesylate (N=144) | Normal Saline (N=147)
Arrhythmia (Cardiac disorders) | 11 (12) | 11 (13)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Colour blindness (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Gaze palsy (Eye disorders) | 1 (1) | 0 (0)
Pupils unequal (Eye disorders) | 1 (1) | 2 (2)
Scleral oedema (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (13) | 6 (6)
Chest pain (General disorders) | 3 (3) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 2 (2) | 5 (6)
Infusion site pain (General disorders) | 2 (2) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 17 (17) | 16 (17)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 18 (18) | 22 (22)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Anaemia (Investigations) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 4 (4) | 6 (6)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 2 (2)
Cardiac enzymes increased (Investigations) | 1 (1) | 2 (2)
Coagulopathy (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 4 (4)
Hyperglycaemia (Investigations) | 7 (7) | 7 (7)
Hypernatraemia (Investigations) | 5 (5) | 1 (1)
Hyperphosphataemia (Investigations) | 1 (1) | 0 (0)
Hypoalbuminaemia (Investigations) | 0 (0) | 1 (1)
Hypocalcaemia (Investigations) | 3 (3) | 3 (3)
Hypokalaemia (Investigations) | 11 (11) | 4 (4)
Hypomagnesaemia (Investigations) | 2 (2) | 2 (2)
Hyponatraemia (Investigations) | 5 (5) | 5 (5)
Hypophosphataemia (Investigations) | 7 (7) | 4 (4)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (2)
Leukocytosis (Investigations) | 5 (5) | 5 (5)
Monocyte count (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Pyuria (Investigations) | 1 (1) | 0 (0)
Rubulavirus test positive (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Brain midline shift (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral hematoma expansion (Nervous system disorders) | 1 (1) | 3 (3)
Convulsion (Nervous system disorders) | 4 (4) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 8 (8)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 5 (5)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 4 (5)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope/Presyncope (Nervous system disorders) | 1 (1) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 13 (15) | 8 (9)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 7 (7) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 9 (9)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 8 (8) | 7 (7)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 6 (6) | 6 (7)
Neurogenic shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-05-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT02175225/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT02175225/SAP_001.pdf